CLINICAL TRIAL: NCT03198286
Title: A Pilot Study of the Clinical Implementation of the Carevive Survivor Care Planning System
Brief Title: Carevive Survivor Care Planning System in Improving Quality of Life in Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 15P.046; JT 7206 (Other: JeffTrial Number)
Record Dates: First submitted 2017-05-19; First posted 2017-06-26 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Stage I Breast Cancer; Stage I Cervical Cancer; Stage I Ovarian Cancer; Stage I Uterine Corpus Cancer; Stage IA Breast Cancer; Stage IA Cervical Cancer; Stage IA Ovarian Cancer; Stage IA Uterine Corpus Cancer; Stage IB Breast Cancer; Stage IB Cervical Cancer; Stage IB Ovarian Cancer; Stage IB Uterine Corpus Cancer; Stage IC Ovarian Cancer; Stage II Breast Cancer; Stage II Cervical Cancer; Stage II Ovarian Cancer; Stage II Uterine Corpus Cancer; Stage IIA Breast Cancer; Stage IIA Cervical Cancer; Stage IIA Ovarian Cancer; Stage IIB Breast Cancer; Stage IIB Cervical Cancer; Stage IIB Ovarian Cancer; Stage IIC Ovarian Cancer; Stage III Breast Cancer; Stage III Cervical Cancer; Stage III Ovarian Cancer; Stage III Uterine Corpus Cancer; Stage IIIA Breast Cancer; Stage IIIA Cervical Cancer; Stage IIIA Ovarian Cancer; Stage IIIA Uterine Corpus Cancer; Stage IIIB Breast Cancer; Stage IIIB Cervical Cancer; Stage IIIB Ovarian Cancer; Stage IIIB Uterine Corpus Cancer; Stage IIIC Breast Cancer; Stage IIIC Ovarian Cancer; Stage IIIC Uterine Corpus Cancer
MeSH Terms: conditions — Breast Neoplasms; Uterine Cervical Neoplasms; Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive care (survivor care plan, survey) (Experimental): Patients receive a customized treatment summary and survivor care plan via the Carevive Survivor Care Planning System and review it during their follow-up visit. Patients also complete a survey on a tablet computer over 10-20 minutes before and after their follow-up visit.
  Interventions: Other: Informational Intervention

INTERVENTIONS:
Other: Informational Intervention — Receive treatment summary and survivor care plan

SUMMARY:
This pilot clinical trial studies how well the Carevive Survivor Care Planning System works in improving quality of life in breast cancer survivors. A personalized survivor care plan includes a summary of a patient's cancer treatment and a customized survivor care plan and may provide beneficial information and resources.

DETAILED DESCRIPTION:
PRIMARY OBJECTIES:

I. To evaluate the feasibility of using the Carevive Survivor Care Planning System (SCPS) during the follow-up visit for breast oncology survivors treated in a university cancer center or a community medical center.

II. To evaluate survivors' perceptions of the usability of the Carevive technology.

III. To evaluate their perceptions of the acceptability (perception of benefit) of the treatment summary and survivor care plan.

SECONDARY OBJECTIVES:

I. Examine the psychometrics of surveys developed for this research. II. Compare participants' perceptions of the care received under the Carevive system with clinician documentation.

III. Compare clinician documentation of care received by this sample with documentation of care provided for historical controls at each site.

ELIGIBILITY:
Inclusion Criteria:

* Prospective study: completed primary treatment for breast malignancies; receive survivorship care at Thomas Jefferson University (TJU) or Reading Health System (RHS)
* Prospective study: individuals will have pathologically confirmed breast cancer (stages I-III)
* Prospective study: Able to understand and read English
* Prospective study: Physically capable of using a tablet computer (no severe visual, hearing, or hand motor deficits)
* Retrospective chart review: Individuals will have pathologically confirmed breast cancer or gynecological (GYN) malignancies including uterine, ovarian, or cervical cancers, stages I-III; treated in the previous two years (2013-2014)

Exclusion Criteria:

* Women who are pregnant
* Vulnerable populations: cognitively impaired; prisoners; terminally ill; elderly and infirm; drug addicts

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2015-08-01 (Actual); Study Completion 2016-10-31 (Actual)

PRIMARY OUTCOMES:
Standard deviation will calculated to identify low-score items indicating problems that need to be addressed. | Up to 1 year
  Feasibility information will be auto-generated by the Carevive system.
Patient reported knowledge and confidence as measured by the Knowledge and Confidence Survey | Up to 1 month
  Survivor reported outcomes will be evaluated.
Patient reported activation as measured by the Patient Activation Survey | Up to 1 month
  Survivor reported outcomes will be evaluated.
Patient reported health behavior as measured by the Health Behavior Survey | Up to 1 month
  Survivor reported outcomes will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Barsevick, PhD, Principal Investigator — Sidney Kimmel Cancer Center at Thomas Jefferson University
Locations (2):
- United States (2):
  - Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania
  - Reading Hospital, Reading, Pennsylvania

REFERENCES:
- See also: Sidney Kimmel Cancer Center — http://www.kimmelcancercenter.org
- See also: Thomas Jefferson University Hospital — http://hospitals.jefferson.edu/